CLINICAL TRIAL: NCT01832155
Title: A Pilot Study Testing a Hatha Yoga Exercise Program in Older Women With Knee Osteoarthritis
Brief Title: Yoga for Managing Knee Osteoarthritis in Older Women: a Feasibility Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: The John A. Hartford Foundation (Other); Midwest Nursing Center Consortium Research Network (Network); St. Catherine University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 1101M95449
Record Dates: First submitted 2013-04-04; First posted 2013-04-15 (Estimated); Results first posted 2014-03-04 (Estimated); Last update posted 2019-11-01 (Actual); Status verified 2019-10

CONDITIONS: Osteoarthritis, Knee; Quality of Life; Poor Quality Sleep; Physical Impairment
Keywords: Yoga; Knee osteoarthritis; Symptom management; Older women; Pain; Stiffness; Physical function); Physical function of the lower extremities; Quality of sleep; Quality of life
MeSH Terms: conditions — Osteoarthritis, Knee; Pain; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- yoga intervention (Experimental): The yoga intervention received eight 60 minute weekly Hatha yoga intervention classes and asked to practice additional 30 minute yoga per day at home.
  Interventions: Behavioral: Hatha yoga
- wait list control (Other): The wait list control group received the same 8-week Hatha yoga intervention involving group and home-based exercise sessions after the yoga intervention group completed the intervention at the end of 8 weeks.
  Interventions: Behavioral: Hatha Yoga

INTERVENTIONS:
Behavioral: Hatha yoga — Hatha yoga poses that were specifically designed by a group of yoga experts for older adults with knee osteoarthritis. Program included physical poses and sequence that focus on strengthening the lower extremities, and relaxation techniques.
  Arms: yoga intervention
Behavioral: Hatha Yoga — The same intervention was provided to the wait-list control group at the end of 8 weeks when the intervention completed their intervention classes.
  Arms: wait list control

SUMMARY:
The study hypothesized that it is feasible and safe to use Hatha yoga in older women with knee osteoarthritis (OA), and practicing Hatha yoga regularly will help reduce pain and stiffness, enhance physical function, and improve quality of sleep and quality of life in older women with knee OA.

DETAILED DESCRIPTION:
1. Potential participants were initially screened via telephone by a trained research assistant for eligibility which was based on the following inclusion criteria:

   1. community-dwelling women aged 65 years or over;
   2. had a symptomatic OA of knee diagnosis for at least 6 months;
   3. had no previous training in any form of yoga; and
   4. were not currently participating in a supervised exercise program.
2. Once initial screening eligibility was established, the individual was seen at home to confirm:

   1. the presence of knee OA symptoms using the Clinical Criteria for the Classification of Idiopathic OA of the Knee developed by the American College of Rheumatology.
   2. Cognitively intact using the Short Portable Mental Status Questionnaire (SPMSQ).
3. Exclusion criteria included:

   * symptoms of joint locking;
   * instability indicated by chronic use of a knee brace, cane, walker, or wheelchair;
   * a corticosteroid injection in the symptomatic joint within three months of study entry;
   * a hyaluronic acid injection in the symptomatic joint within six months of study entry;
   * a history of knee surgery within the last two years or a joint replacement at any point;
   * individuals who had self-reported significant medical comorbidities that might preclude exercise participation such as: a) uncontrolled high blood pressure or existing heart condition; and b) other comorbid condition with overlapping symptoms (i.e. fibromyalgia, rheumatoid arthritis);
   * individuals who had medication changes for arthritis symptoms were permitted to remain in the trial; however, these changes were monitored.
4. Primary outcome measures included:

   - OA symptoms (e.g., pain, stiffness and physical function) were assessed using the Western Ontario and McMaster Universities OA Index scale (LK scale 3.1) (WOMAC) and a single question that asked about the number of pain medications used per day.
   * WOMAC scale contains 24 items divided into 3 subscales: Pain (5 items), Stiffness (2 items), and Physical Function (17 items). The 5-point Likert Scale uses the following descriptors for all items: none, mild moderate, severe, and extreme. These correspond to an ordinal scale of 0-4. The scores are summed for items in each subscale, with possible ranges as follows: pain=0-20, stiffness=0-8, physical function=0-68. A total WOMAC score is created by summing the items for all three subscales. Higher values represent a worse OA symptom.
5. Secondary outcome measures included:

   * physical performance of the LE which was assessed using the Short Physical Performance Battery (SPPB) developed by the National Institute on Aging. The test consists of three components: repeated chair stands, balance, and timed 8" walk. Each subscale 0 (worst performance) to 12 (best performance).
   * BMI in kg/m^2 was calculated using the participant's weight and height.
   * Quality of sleep was evaluated using the Pittsburgh Sleep Quality Index (PSQI). A score of ≥ 5 on the PSQI total scale, which is computed as a sum of the seven subscales (e.g., sleep quality, sleep latency, sleep duration, sleep disturbance, sleep efficiency, and use sleep medication) is associated with clinically significant sleep disruptions, including insomnia and major mood disorders.
   * The self-perceived quality of life was assessed using the Short Form Health Survey (SF-12) which measures a total of 8 health domains: 4 physical and 4 mental component summary scales. Physical Health (physical functioning, role-physical, bodily pain, and general health)and Mental Health (vitality, social functioning, role-emotional, and mental health) Composite Scores (PCS & MCS) are computed using the scores of twelve questions and range from 0 to 100, where a zero score indicates the lowest level of health measured by the scales and 100 indicates the highest level of health. The Cantril Self-Anchoring Ladder that measures both "current" and "in 5 years" using steps from 0 to 10, where "0" represents the worst possible life and "10" represents the best possible life.
6. Feasibility measures: Feasibility was measured by eligibility, recruitment, and retention rates.

   * The average number of yoga class attendance and minutes of home practice were used to measure the retention and adherence rates.
   * Acceptability was evaluated by the participants' perceived difficulty of the yoga class and level of enjoyment.
   * Perceived level of difficulty and enjoyment were rated by participants after completing the yoga program on two different scales of 1 - 10 where 10 represents "extremely difficult" and "most enjoyable", respectively.
   * Safety was assessed by recording the frequency of injuries that occur during group and home-based exercise sessions.
7. Demographic information (e.g., age, race/ethnic background, education level, annual household income, marital status, living arrangement, and type of insurance), and comorbidities were collected from all participants.

ELIGIBILITY:
Inclusion Criteria:

* community-dwelling women aged 65 years or over
* had a symptomatic OA of knee diagnosis for at least 6 months
* had no previous training in any form of yoga; and
* were not currently participating in a supervised exercise program
* cognitively intact

Exclusion Criteria:

* symptoms of joint locking;
* instability indicated by chronic use of a knee brace, cane, walker, or wheelchair;
* a corticosteroid injection in the symptomatic joint within three months of study entry;
* a hyaluronic acid injection in the symptomatic joint within six months of study entry;
* a history of knee surgery within the last two years or a joint replacement at any point;
* individuals who had self-reported significant medical comorbidities that might preclude exercise participation such as: a) uncontrolled high blood pressure or existing heart condition; and b) other comorbid condition with overlapping symptoms (i.e. fibromyalgia, rheumatoid arthritis) were also be excluded.

Ages: 65 Years to 86 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 36 (Actual)
Dates: Start 2011-01; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Corjena K Cheung, PhD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

REFERENCES:
- [Derived] Cheung C, Wyman JF, Resnick B, Savik K. Yoga for managing knee osteoarthritis in older women: a pilot randomized controlled trial. BMC Complement Altern Med. 2014 May 18;14:160. doi: 10.1186/1472-6882-14-160. PMID 24886638

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment took 9 months through placing flyers in various community centers; distributing press releases to the University's Alumnae Newsletter, community newsletters and newspapers; presenting health talks at community senior programs; and accessing the data base and mailing invitation letters out to patients from the University Clinic.
Pre-assignment Details: No significant events and approaches for the overall study following participant enrollment/prior to group assignment.
Groups:
- Wait List Control: The wait list control group received the same 8-week Hatha yoga intervention involving group and home-based exercise sessions after the yoga intervention group completed the intervention at the end of 8 weeks.
  Hatha Yoga : The same intervention was provided to the wait-list control group at the end of 8 weeks when the intervention completed their intervention classes.
- Yoga Intervention: The yoga intervention received eight 60 minute weekly Hatha yoga intervention classes and asked to practice additional 30 minute yoga per day at home.
  Hatha yoga : Hatha yoga poses that were specifically designed by a group of yoga experts for older adults with knee osteoarthritis. Program included physical poses and sequence that focus on strengthening the lower extremities, and relaxation techniques.
Period: Beginning of Study: Baseline at 0 Week
Arm/Group | Wait List Control | Yoga Intervention
Started | 18 | 18
Completed | 17 | 18
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Period: Mid-point of Study: 0 - 4 Weeks
Arm/Group | Wait List Control | Yoga Intervention
Started | 17 | 18
Completed | 16 | 18
Not Completed | 1 | 0
Not completed — Protocol Violation | 1 | 0
Period: End of Study: 4 - 8 Weeks
Arm/Group | Wait List Control | Yoga Intervention
Started | 16 | 18
Completed | 16 | 18
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Wait List Control | Yoga Intervention | Total
Number analyzed (Participants) | 18 | 18 | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 18 | 18 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.9 (6.0) | 71.9 (5.4) | 71.9 (5.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 18 | 36
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 18 | 18 | 36

OUTCOME MEASURES:

1. Primary Outcome: Absolute Value of OA Symptoms at 8 Weeks
Description: Primary outcome measures included: OA symptoms (pain, stiffness and function) were assessed using the Western Ontario and McMaster Universities OA Index scale (LK scale 3.1)(WOMAC). The WOMAC measures five items for pain (score range 0-20), two for stiffness (score range 0-8), and 17 for functional limitation (score range 0-68). A total WOMAC score is created by summing the items for all three subscales resulting in a possible score of 0 - 96. Higher scores on the WOMAC indicate worse pain, stiffness, and functional limitations.
Time Frame: 8 weeks
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Wait List Control | Yoga Intervention
Number analyzed (Participants) | 18 | 18
units on a scale | 39.3 (3.0) | 31.0 (3.0)

2. Secondary Outcome: Absolute Value of Physical Performance of the Lower Extremities (LE) at 8 Weeks
Description: Secondary outcome measures included physical performance of the LE which was assessed using the Short Physical Performance Battery (SPPB) developed by the National Institute on Aging. The test consists of three components: repeated chair stands (4 points), balance (4 points), and timed 8" walk (4 points). A maximum score of 12 points can be achieved. Higher values indicate better physical functions.
Time Frame: 8 weeks
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Wait List Control | Yoga Intervention
Number analyzed (Participants) | 18 | 18
units on a scale | 9.0 (.37) | 10.0 (.37)

3. Secondary Outcome: Absolute Value of Quality of Sleep at 8 Weeks
Description: Pittsburgh Sleep Quality Index (PSQI) was used to measure quality of sleep. The PSQI is a 19-item self-rated questionnaire for evaluating subjective sleep quality over the previous month. The 19 questions are combined into 7 clinically-derived component scores, each weighted equally from 0-3 whereby 3 reflects the negative extreme on the Likert Scale. The 7 component scores are added to obtain a global score ranging from 0-21, with higher scores indicating worse sleep quality. A global score of ≥ 5 on the PSQI total scale, which is computed as a sum of the seven subscales (e.g., sleep quality, sleep latency, sleep duration, sleep disturbance, sleep efficiency, and use sleep medication) is associated with clinically significant sleep disruptions, including insomnia and major mood disorders.
Time Frame: 8 weeks
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Wait List Control | Yoga Intervention
Number analyzed (Participants) | 18 | 18
units on a scale | 6.1 (.52) | 5.0 (.52)

4. Secondary Outcome: Absolute Value of Quality of Life at 8 Weeks
Description: The self-perceived quality of life was assessed using the Short Form Health Survey (SF-12) which measures a total of 8 health domains: 4 physical and 4 mental component summary scales. Physical Health (physical functioning, role-physical, bodily pain, and general health)and Mental Health (vitality, social functioning, role-emotional, and mental health) Composite Scores (PCS & MCS) are computed using the scores of twelve questions and range from 0 to 100, where a zero score indicates the lowest level of health measured by the scales and 100 indicates the highest level of health. The Cantril Self-Anchoring Ladder that measures both "current" and "in 5 years" using steps from 0 to 10, where "0" represents the worst possible life and "10" represents the best possible life.
Time Frame: 8 weeks
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Wait List Control | Yoga Intervention
Number analyzed (Participants) | 18 | 18
units on a scale
  SF12 MCS | 51.7 (1.2) | 49.7 (1.2)
  SF12 PCS | 38.7 (1.0) | 38.0 (.98)
  Cantril Ladder current | 7.7 (.37) | 7.5 (.37)
  Cantril Ladder in 5 years | 7.8 (.32) | 7.2 (.32)

5. Secondary Outcome: Absolute Value of BMI at 8 Weeks
Description: BMI was calculated using the participant's weight and height, kg/m^2.
Time Frame: 8 weeks
Measure: Mean (Standard Error); unit: kg/m^2
Arm/Group | Wait List Control | Yoga Intervention
Number analyzed (Participants) | 18 | 18
kg/m^2 | 28.9 (.16) | 28.7 (.16)

6. Other Pre Specified Outcome: Feasibility Measures - Retention
Description: Feasibility was measured by the retention rate during the 8 weeks program. Data from both intervention and wait-list control (during their treatment period) groups were collected. Participants' class attendance (average number of classes attended) was evaluated.
Time Frame: 8 weeks
Measure: Mean (Full Range); unit: classes
Groups:
- Class Rentention: The yoga intervention received eight 60 minute weekly Hatha yoga intervention classes and asked to practice additional 30 minute yoga per day at home.
  Hatha yoga : Hatha yoga poses that were specifically designed by a group of yoga experts for older adults with knee osteoarthritis. Program included physical poses and sequence that focus on strengthening the lower extremities, and relaxation techniques.
Arm/Group | Class Rentention
Number analyzed (Participants) | 35
classes | 6 [1 to 8]

7. Other Pre Specified Outcome: Feasibility Measures - Adherence
Description: Feasibility was also measured by the home practice adherence rate during the 8 weeks program. Data from both intervention and wait-list control (during their treatment period) groups were collected. Home yoga practice adherence was determined by participants' report of the average number of minutes of yoga practiced at home.
Time Frame: 8 Weeks
Measure: Mean (Full Range); unit: minutes/week
Groups:
- All Participants: The yoga intervention received eight 60 minute weekly Hatha yoga intervention classes and asked to practice additional 30 minute yoga per day at home.
  Hatha yoga : Hatha yoga poses that were specifically designed by a group of yoga experts for older adults with knee osteoarthritis. Program included physical poses and sequence that focus on strengthening the lower extremities, and relaxation techniques.
Arm/Group | All Participants
Number analyzed (Participants) | 33
minutes/week | 112 [21 to 190]

8. Other Pre Specified Outcome: Feasibility Measure - Acceptability
Description: Acceptability was evaluated by the participants' perceived difficulty of the yoga class and level of enjoyment. Upon completion of the yoga program, perceived level of program difficulty was rated by participants using a scale of 1 - 10 where 10 represents "extremely difficult" and a scale of 1 - 10 where 10 represents "most enjoyable" was used to measure perceived level of program enjoyment. Data from both intervention and wait-list control (during the intervention period) groups were collected.
Time Frame: 8 weeks
Measure: Mean (Full Range); unit: units on a scale
Groups:
- About the Yoga Intervention: The yoga intervention received eight 60 minute weekly Hatha yoga intervention classes and asked to practice additional 30 minute yoga per day at home.
  Hatha yoga : Hatha yoga poses that were specifically designed by a group of yoga experts for older adults with knee osteoarthritis. Program included physical poses and sequence that focus on strengthening the lower extremities, and relaxation techniques.
Arm/Group | About the Yoga Intervention
Number analyzed (Participants) | 35
units on a scale
  Level of difficulty | 4 [0 to 9]
  level of enjoyment | 9 [5 to 10]

9. Other Pre Specified Outcome: Feasibility Measure - Safety
Description: Safety was assessed by measuring the frequency of yoga related injuries that occur from group or home-based exercise sessions during the active treatment periods.
Time Frame: 8 weeks
Measure: Number; unit: injuries
Groups:
- Both Groups During Yoga Intervention: The yoga intervention received eight 60 minute weekly Hatha yoga intervention classes and asked to practice additional 30 minute yoga per day at home.
  Hatha yoga : Hatha yoga poses that were specifically designed by a group of yoga experts for older adults with knee osteoarthritis. Program included physical poses and sequence that focus on strengthening the lower extremities, and relaxation techniques.
Arm/Group | Both Groups During Yoga Intervention
Number analyzed (Participants) | 36
injuries
  Number of yoga related injuries in class | 0
  Number of yoga home practice related injuries | 0

10. Primary Outcome: Absolute Value of OA Pain at 8 Weeks
Description: A single question that asked about the number of pain medications used per day for knee OA was also used to measure OA pain status.
Time Frame: 8 weeks
Measure: Mean (Standard Error); unit: Number of pain medication/day
Groups:
- Wait-list Control Group: Participants in the control group received the same Hatha yoga program at the end of 8 weeks when the intervention group completed their intervention classes.
- Yoga Intervention Group: The yoga intervention received eight 60 minute weekly Hatha yoga intervention classes and asked to practice additional 30 minute yoga per day at home.
  Hatha yoga : Hatha yoga poses that were specifically designed by a group of yoga experts for older adults with knee osteoarthritis. Program included physical poses and sequence that focus on strengthening the lower extremities, and relaxation techniques.
Arm/Group | Wait-list Control Group | Yoga Intervention Group
Number analyzed (Participants) | 18 | 18
Number of pain medication/day | 1 (1.4) | 1 (1.3)

11. Other Pre Specified Outcome: Feasibility Measure - Recruitment
Description: The number of months it took to recruit 36 participants.
Time Frame: 9 months
Measure: Number; unit: months
Arm/Group | All Participants
Number analyzed (Participants) | 36
months | 9

ADVERSE EVENTS:
Arm/Group | Wait List Control | Yoga Intervention
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/18
Other Adverse Events (participants affected / at risk) | 0/18 | 0/18

LIMITATIONS AND CAVEATS:
Limitations: Small sample size without blinding. Strengths: Randomized controlled design, data collection at multiple time points and the use of a yoga expert panel to design the yoga program specifically for older women with knee osteoarthritis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes